CLINICAL TRIAL: NCT03959943
Title: Sensory Recovery of the Breast Following Innervated and Non-innervated Lateral Thigh Perforator (LTP) Flap Breast Reconstructions
Brief Title: Nerve Coaptation in LTP Flap Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Rene van der Hulst, Head of the Plastic Surgery department, Maastricht University Medical Center
Other Study IDs: METC16-4-147
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; LTP flap; Sensory recovery; Breast sensation; Nerve coaptation
MeSH Terms: conditions — Breast Neoplasms | interventions — Nerve Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Innervated LTP flaps: Patients in this group underwent immediate or delayed, unilateral or bilateral lateral thigh perforator (LTP) flap breast reconstruction with additional sensory nerve coaptation.
  Interventions: Procedure: Sensory nerve coaptation
- Non-innervated LTP flaps: Patients in this group underwent immediate or delayed, unilateral or bilateral lateral thigh perforator (LTP) flap breast reconstruction without sensory nerve coaptation.

INTERVENTIONS:
Procedure: Sensory nerve coaptation — A recipient sensory nerve branch of the lateral cutaneous femoral nerve (LCFN) was reattached to a donor nerve in the chest area. The anterior cutaneous branch of the second or third intercostal nerve was used as the donor nerve. Direct, end-to-end nerve coaptation was performed.
  Other Names: Neurotization; Reinnervation
  Groups: Innervated LTP flaps

SUMMARY:
The sensory recovery of the breast remains an undervalued aspect of breast reconstruction and surgical reinnervation is not regarded as a priority by most reconstructive surgeons. A prospective study was conducted of all patients who underwent either innervated or non-innervated lateral thigh perforator (LTP) flap breast reconstruction in Maastricht University Medical Center and returned for follow-up between February 2016 and April 2019. Semmes-Weinstein monofilaments were used for sensory testing of the breast.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older
* Unilateral or bilateral LTP flap breast reconstruction
* Returned for follow-up between February 2016 and April 2019
* Informed consent

Exclusion Criteria:

* In case of a total flap loss
* Flaps that required a take-back
* Follow-up less than six months postoperatively

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients of 18 years or older.
Study Population: In this prospective study, patients who underwent an innervated or non-innervated LTP flap breast reconstruction between December 2014 and August 2018 at Maastricht University Medical Center in the Netherlands were included if they returned for follow-up between February 2016 and April 2019.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The sensory recovery of the reconstructed breast as assessed by Semmes-Weinstein monofilaments | Through study completion up to 27 months postoperatively
  The sensory recovery of the breast to touch was tested at different follow-up moments after the initial surgery. Semmes-Weinstein monofilaments were used for sensory testing. Nine areas of the breast, indicating native skin and flap skin, were tested. Mean monofilament values were calculated for each area and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: René van der Hulst, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No